CLINICAL TRIAL: NCT07202884
Title: A Master Protocol to Investigate the Efficacy and Safety of Orforglipron Tablet Once Daily Compared With Placebo in Female Participants With Stress Urinary Incontinence Who Have Obesity or Overweight
Brief Title: A Study of Orforglipron in Female Participants With Stress Urinary Incontinence Who Have Obesity or Overweight
Acronym: RESTRAIN-SUI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27672; 2025-522514-23-00 (EU CTIS Number); J2A-MC-GZPS (Other: Eli Lilly and Company); J2A-MC-GZS1 (Other: Eli Lilly and Company); J2A-MC-GZS2 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orforglipron (GZS1) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (GZS1) (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo
- Orforglipron (GZS2) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (GZS2) (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron (GZS1); Orforglipron (GZS2)
Drug: Placebo — Administered orally
  Arms: Placebo (GZS1); Placebo (GZS2)

SUMMARY:
The GZPS master protocol will support two independent studies, J2A-MC-GZS1 and J2A-MC-GZS2. Each study will see how well and safely orforglipron works in adult female participants with stress urinary incontinence (SUI) who have obesity or overweight. SUI is leaking urine during movement or activity such as coughing or exercising. Participation in the study will last about 58 weeks from screening to safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of 27 kilograms per square meter (kg/m2) or higher at screening
* Have a diagnosis of stress urinary incontinence

Exclusion Criteria:

* Have had urinary incontinence surgery
* Have recently received onabotulinumtoxin A (Botox) bladder injections or currently taking medications for urinary incontinence
* Have given birth within one year of screening
* Have had a change in body weight of more than 11 pounds within 90 days prior to screening
* Have used any anti-obesity medication or alternative weight loss remedies within 180 days prior to screening
* Have type 1 diabetes, type 2 diabetes, or any other type of diabetes
* Have had a cardiovascular health condition within 90 days prior to screening
* Are pregnant, intending to be pregnant, breastfeeding, or intending to breastfeed for the duration of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Incontinence Episode Frequency (IEF) | Baseline, Week 52

SECONDARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 52
Change from Baseline in Urinary Incontinence-Specific Quality of Life | Baseline, Week 52
Change from Baseline in Number of Continence Pad (CAPD) Used Per Week | Baseline, Week 52
Change from Baseline in Patient Global Impression of Condition | Baseline, Week 52
Percent Change from Baseline in Total Cholesterol | Baseline, Week 52
Change from Baseline in Waist Circumference | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (133):
- United States (21):
  - University of Alabama -The Kirklin Clinic, Birmingham, Alabama
  - AMR Clinical, Mobile, Alabama
  - Urologic Surgeons of Arizona, Mesa, Arizona
  - Matrix Clinical Research, Los Angeles, California
  - Alarcon Urology Center, Montebello, California
  - Prestige Medical Group, Tustin, California
  - Colorado Clinical Research, Lakewood, Colorado
  - AMR Clinical, Fort Myers, Florida
  - Altus Research, Lake Worth, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Emerald Coast OBGYN Clinical Research, Panama City, Florida
  - Teak Research Consults, Lawrenceville, Georgia
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - OB/GYN Associates of Erie, Erie, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Next Level Urgent Care, Houston, Texas
  - Innovative Medical Research of Texas, Houston, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Clinical Research Center, Seattle, Washington
- Canada (8):
  - OCT Research ULC, Kelowna
  - Kelowna Health and Memory Centre, Kelowna
  - Alpha Recherche Clinique - Lévis, Lévis
  - The Fe/Male Health Centre, Oakville
  - Alpha Recherche Clinique, Québec
  - ALPHA Recherche Clinique, Québec
  - CaRe Clinic, Red Deer
  - Sunnybrook Research Institute, Toronto
- China (20):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Chengdu Women and Children Center Hospital, Chengdu
  - 2nd Affiliated Hospital Chongqing Medical University, Chongqing
  - Zhujiang Hospital, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Second Affiliated hospital of Anhui Medical University, Hefei
  - Gansu Provincial Hospital, Lanzhou
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Ningbo First Hospital, Ningbo
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai
  - Peking University Shenzhen Hospital, Shenzhen
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated hospital of Xiamen University, Xiamen
  - General Hospital of Ningxia Medical University, Yinchuan
- Czechia (9):
  - Afimed - Urologicka ambulance, Benešov
  - Gynekologie Šottner, Brno
  - Centrum Panevniho Dna, Karlovy Vary
  - Kestr-gyn, Náchod
  - G-CENTRUM Olomouc, Olomouc
  - NEUMED gynekologická ambulance, Olomouc
  - GYNORD plus, Ostrava
  - Gyncare, Pilsen
  - Nestátní zdravotnické zařízení GONA, Prague
- India (15):
  - Devasya Superspeciality Kidney & Multispeciality Hospitals, Ahmedabad
  - Apollo Hospitals Ahmedabad, Ahmedabad
  - KLES Dr. Prabhakar Kore Hospital & M.R.C, Belagavi
  - Belagavi Institute of Medical Sciences - Belagavi, Belgavi
  - All India Institute of Medical Sciences, Bhubaneswar
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Apollo Hospitals - Chennai, Chennai
  - Malla Reddy Narayana Multispeciality Hospital, Hyderabad
  - Ketki Nursing Home & Urology Hospital, Nagpur
  - Sir Ganga Ram Hospital, New Delhi
  - Lifepoint Multispeciality Hospital, Pune
  - All India Institute of Medical Sciences, Raipur
  - All India Institute of Medical Sciences - Rishikesh, Rishikesh
  - Surat Institute of Digestive Sciences Hospitals, Surat
  - Banaras Hindu University, Varanasi
- Japan (17):
  - Hasegawa Hospital - Arakawa, Arakawa City
  - Takasu Nephrology and Urology Clinic, Chiba
  - Yotsuya Medical Cube, Chiyoda City
  - St. Luke's International Hospital, Chūōku
  - Mito Medical Center, Higashiibaraki
  - Nihon University Itabashi Hospital, Itabashiku
  - Kokura Memorial Hospital, Kitakyushu
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Koujunkai Daido Clinic, Nagoya
  - Women's Clinic LUNA NEXT STAGE, Naka-ku, Yokohama-Shi
  - Nakazawa Nephrology and Urology Clinic, Nonoichi
  - Miyabi Urogyne Clinic, Okayama
  - Yukigaya Urology Clinic, Ōta-ku
  - Kashiwazaki Obstetrics and Gynecology Clinic, Saitama-shi
  - Izumi Chuo Hospital, Sendai
  - Toride Urology Clinic, Toride
  - Tsukuba Urocare Clinic, Tsukuba
- Mexico (13):
  - Medical Center Metas, Chihuahua City
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C., Ciudad Madero
  - Health Pharma Querétaro, Juriquilla
  - Centro de Oncología de Precisión - Mexico City, Mexico City
  - RM Pharma Specialists - Unidad Especializada en Datos, Mexico City
  - Quemex Medical and Research, Mexico City
  - Medical Care and Research SA de CV, Mérida
  - Clinstile, S.A. de C.V., México
  - Jose Gerardo Garza Leal, Monterrey
  - Centro de investigación y control metabólico, Monterrey
  - Centro de Investigacion Clinica Chapultepec, Morelia
  - Medimanage Research, Tlalpan
- Poland (6):
  - IN VIVO, Bydgoszcz
  - AIDPORT Sp. z o.o., Skórzewo
  - Centrum Medyczne Euromedis, Szczecin
  - Medical Concierge Centrum Medyczne, Warsaw
  - Centrum Medyczne Ginemedica, Wroclaw
  - EMC Instytut Medyczny SA, Wroclaw
- Romania (17):
  - Centrul Medical Unirea, Brasov
  - Spitalul Clinic Judetean de Urgenta (Brasov), Brasov
  - Spitalul Clinic de Nefrologie Doctor Carol Davila, Bucharest
  - Spitalul Universitar de Urgenta Militar Central Dr. Carol Davila, Bucharest
  - Delta Health Care, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul de Urgenta al Ministerului Administratiei si Internelor "Prof. Dr. Dimitrie Gerota", Bucharest
  - Spitalul Clinic Județean de Urgență Ilfov, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Gnosis Evomed S.R.L., Bucharest
  - Spitalul Clinic Profesor Doctor Theodor Burghele, Bucharest
  - Spitalul Clinic Județean de Urgență, Craiova
  - Spitalul Clinic Judetean De Urgenta Bihor, Oradea
  - Clinica Polisano, Sibiu
  - Polaris Medical SA, Suceagu
  - S.C. Materna Care S.R.L., Timișoara
  - Spitalul Clinic Judeţean de Urgenţă Pius Brînzeu Timişoara, Timișoara
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si
  - Pusan National University Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Kyungpook National University Hospital, Junggu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Orforglipron in Female Participants With Stress Urinary Incontinence Who Have Obesity or Overweight (RESTRAIN-SUI) — https://trials.lilly.com/en-US/trial/658355